CLINICAL TRIAL: NCT05850572
Title: A Prospective, Double-blind, Randomized Controlled Trial of FMT Combined With Antidepressants to Improve the Efficacy in Patients With Depressive Disorder
Brief Title: A Study of the Efficacy of Fecal Microbiota Transplantation(FMT) in the Treatment of Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 82022023-1; 2021GXLH-Z-083-1 (Other Grant/Funding Number: Key Research and Development Plan of Shaanxi Province)
Record Dates: First submitted 2023-04-12; First posted 2023-05-09 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbiota transplantation(FMT) (Experimental): Subjects will receive FMT capsules (10^12 CFU/capsule) in addition to their usual antidepressant treatment. Subjects will continue to receive FMT capsules for 8 weeks. New SSRI antidepressants (fluoxetine, citalopram, escitalopram, sertraline, paroxetine, and fluvoxamine) recommended by current treatment guidelines can be used during this period, and the effective therapeutic dose of the drugs can be added within 1 week.
  Interventions: Drug: Fecal microbiota transplantation(FMT)
- Placebo (Placebo Comparator): Participants will receive a placebo capsule with the same color, appearance, and smell as the FMT capsule, in addition to their usual antidepressant treatment. Placebo capsules contained the food probiotic Lactobacillus (10^12 CFU per capsule). Subjects will continue to receive placebo capsules for 8 weeks. New SSRI antidepressants (fluoxetine, citalopram, escitalopram, sertraline, paroxetine, and fluvoxamine) recommended by current treatment guidelines can be used during this period, and the effective therapeutic dose of the drugs can be added within 1 week.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fecal microbiota transplantation(FMT) — Subjects will receive FMT capsules (10^12 CFU/capsule) in addition to their usual antidepressant treatment. Subjects will continue to receive FMT capsules for 8 weeks. New SSRI antidepressants (fluoxetine, citalopram, escitalopram, sertraline, paroxetine, and fluvoxamine) recommended by current treatment guidelines can be used during this period, and the effective therapeutic dose of the drugs can be added within 1 week.
  Arms: Fecal microbiota transplantation(FMT)
Other: Placebo — Participants will receive a placebo capsule with the same color, appearance, and smell as the FMT capsule, in addition to their usual antidepressant treatment. Placebo capsules contained the food probiotic Lactobacillus (10^12 CFU per capsule). Subjects will continue to receive placebo capsules for 8 weeks. New SSRI antidepressants (fluoxetine, citalopram, escitalopram, sertraline, paroxetine, and fluvoxamine) recommended by current treatment guidelines can be used during this period, and the effective therapeutic dose of the drugs can be added within 1 week.
  Arms: Placebo

SUMMARY:
Patients with depression were enrolled and randomly divided into two groups, namely FMT combined with antidepressant group and Antidepressant alone group.The former received FMT capsules and antidepressants, and the latter received oral placebo and antidepressants for an 8-week intervention.Before and after intervention, venous blood samples were collected from patients for routine tests such as liver and kidney function to judge the safety of treatment. At the same time, psychological scales were used to evaluate the improvement of patients' depressive symptoms, so as to judge the efficacy and safety of FMT combined with antidepressants.

DETAILED DESCRIPTION:
The main research content of this project is to observe the efficacy and safety of adjuvant FMT capsules in the treatment of depression by recruiting patients with first episode depression and randomly administering FMT combined with antidepressants or placebo combined with antidepressants.

In this study, patients with first episode depression were randomly divided into two groups. The first group was the experimental group, and FMT capsules (10^12 colony forming unit(CFU)/ capsule) were used in addition to conventional antidepressant therapy. The other group, a control group, was given placebo capsules with the same color, look and smell as the FMT capsules in addition to regular antidepressant therapy. Placebo capsules contain Lactobacillus probiotics for food use (10^12 CFU/ capsule). The changes of depressive symptoms and adverse reactions before and after treatment were observed in the two groups to explore the efficacy and safety of FMT capsule in the adjuvant treatment of depression.

The subjects (inpatients) were evaluated for meeting the eligibility requirements for this study according to the pre-specified inclusion and exclusion criteria, and demographic data (age, sex, marital status, educational level, employment, height and weight, smoking and drinking, and other general information as well as questionnaire assessment of eating habits) were collected. Improve laboratory examination (blood routine, liver function, kidney function and lipid), electrocardiogram and scale assessment.

Patients at the end of the screening period were randomly assigned to the experimental and control groups. Subjects will continue to receive FMT capsules or placebo capsules until the end of 8 weeks. During this period, both groups could use new selective serotonin reuptake inhibitors(SSRI)(fluoxetine, citalopram, escitalopram, Sertraline, paroxetine and fluvoxamine) recommended by current treatment guidelines, and the effective therapeutic dose of the drugs was added within 1 week. If, during the 8 weeks of the treatment period, the patient experienced significant fluctuations or severe adverse events that necessitates a change in antidepressant class, the study was terminated.

Benzodiazepines and medications that ameliorate side effects of antidepressants were allowed during the study period. Antipsychotics and mood stabilizers were prohibited. Electronic biofeedback therapy was allowed during the study, and transcranial magnetic stimulation and electroconvulsive non-convulsive therapy were prohibited.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 65 years
* Patients with first-episode depression who met the International Classification of Diseases(ICD)-10 diagnosis of depression
* Hamilton Depression Scale (HAMD) score ≥17
* Informed consent was obtained.

Exclusion Criteria:

* Use of antibiotics within 1 month
* Women are pregnant and lactating
* Patients with severe unstable cardiovascular disease, liver disease, kidney disease, etc
* Patients with malignant tumor or serious systemic disease
* Suffering from other mental disorders such as bipolar disorder, obsessive-compulsive disorder
* It is accompanied by intestinal diseases that seriously damage the intestinal barrier, such as inflammatory bowel disease, Crohn's disease, intestinal tuberculosis, ischemic bowel disease, and radiation enteritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale | At the beginning of treatment
  Hamilton Depression Scale (HAMD) is the most commonly used scale in clinical depression assessment. The minimum and maximum values of HAMD were 0 and 24; Higher scores mean a worse outcome.
Hamilton Depression Scale | At the end of 4 weeks
  Hamilton Depression Scale (HAMD) is the most commonly used scale in clinical depression assessment. The minimum and maximum values of HAMD were 0 and 24; Higher scores mean a worse outcome.
Hamilton Depression Scale | At the end of 8 weeks
  Hamilton Depression Scale (HAMD) is the most commonly used scale in clinical depression assessment. The minimum and maximum values of HAMD were 0 and 24; Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Zhu, professor, Study Director — First Affiliated Hospital Xi'an Jiaotong University